CLINICAL TRIAL: NCT04947228
Title: Supervised Exercise Therapy Using Mobile Health Technology in Patients With Peripheral Arterial Disease: Randomized Controlled Pilot Trial.
Brief Title: Digital Support for Supervised Exercise Therapy in Peripheral Arterial Disease
Acronym: TrackPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Julia Lortz, Assistant Professor, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-8355-BO
Record Dates: First submitted 2021-06-09; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): in addition to the usual therapy, the patients were given access to the trackPAD app
  Interventions: Device: trackPAD
- control group (No Intervention): patients in this group were treated as usual in the clinic without additional interventions.

INTERVENTIONS:
Device: trackPAD — TrackPAD is a smartphone app to provide PAD-specific support for SET
  Arms: intervention group

SUMMARY:
The individual restrictions of daily life for patients with PAD are more important than statistical facts for mortality and morbidity. Intermittent claudication causes a progressive reduction of the pain-free walking distance (PWD) as an expression of a worsening PAD. This decrease in physical capability results in a decline of mental health and relevantly reduces the patients' quality of life (QoL).

Supervised exercise therapy (SET) is a cornerstone in the conservative management of intermittent claudication and extends the PWD. Even though SET is easy to practice and highly cost effective, the adherence to perform SET on a regular base is rather low. The underuse of exercise can be partly explained by the lack of institutional resources, but also by both patients' and physicians' lack of interest in exercise.

Mobile health (mHealth) technologies increase the incentives and provide digital support for patients with PAD on several treatment levels. They might lead to a higher adherence to exercise training and offer new scopes in patient-centered healthcare, but so far studies show opposite results. Because app stores are flooded with health and fitness apps, specific support tools are highly desired by patients with PAD and PAD-specific solutions are missing so far. Based on this background, the investigators developed a smartphone app named TrackPAD to provide PAD-specific support for SET.

The TrackPAD pilot study was designed as a 2-armed randomized controlled trial and included patients with diagnosed and symptomatic PAD. Patients were randomized by the Center for Clinical Studies in Essen using the TENALEA software into 2 groups. The control group included participants with standard care and no further mobile intervention. The intervention group included participants with standard care and additional mHealth-based self-tracking of their physical activity using trackPAD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lower extremity PAD based on (and/or):

  * ABI ≤ 0.9 in at least one legs
  * Invasive or non-invasive imaging of stenotic lower extremity artery disease
  * Endovascular or surgical revascularization of lower extremity artery
* PAD Fontaine Stage IIa/b
* Smartphone with possibility to use TrackPAD: Android ≥ 5.0 or IOS ≥ 11.0
* Written informed consent prior to any study procedures, including a specified follow-up evaluation
* Best-medical treatment in the last 2 months in accordance with standard guidelines

Exclusion Criteria:

* Wheelchair bound, use of walking aid or walking impairment due to another cause than PAD
* Below or above knee amputation
* Acute or critical limb ischemia
* PAD Fontaine Stage I or III / IV
* No German knowledge
* Severe cognitive dysfunction
* Congestive heart failure with NYHA III-IV symptoms
* Active congestive heart failure requiring the initiation or uptitration of diuretic therapy
* Angina pectoris with CCS class 3-4 symptoms or myocardial infarction or stroke in the last 3 months
* Active arrhythmia requiring the initiation or uptitration of anti-arrhythmic therapy
* Severe valve disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
change in 6-minutes walking distance | baseline, 3 months follow-up
  measured via GPS with the trackPAD app

SECONDARY OUTCOMES:
change in physical activity, measured in patients' self-report on how many days a week on average they engage in a physical activity that causes them to sweat or get out of breath, and how many minutes on average they spend doing it. | baseline, 3 months follow-up
  to compare the two groups groups in terms of physical endurance, the self-reported physical activity was recorded
peripheral arterial disease-related quality of life | baseline, 3 months follow-up
  measured with the Peripheral artery disease Quality of Life Questionnaire (PADQOL) questionnaire, a validated PAD-specific questionnaire. Minimum score is 38 and maximum is 228, with higher values indicating a better outcome.
Usability of the TrackPAD app | baseline, 3 months follow-up
  measured with the User version of the Mobile Application Rating Scale (uMars) questionnaire. The uMARS includes 3 factors, namely app quality, app subjective quality and perceived impact. Minimum score of the app quality scale is 4 and the maximum is 20. The App Subjective Quality scale has a minimum of 4 and a maximum of 20, and the Perceived Impact scale has a minimum of 6 and a maximum of 30. Higher values indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lortz, Principal Investigator — University Hospital, Essen
Locations (1):
- Department of Cardiology and Vascular Medicine, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paldan K, Simanovski J, Ullrich G, Steinmetz M, Rammos C, Janosi RA, Moebus S, Rassaf T, Lortz J. Feasibility and Clinical Relevance of a Mobile Intervention Using TrackPAD to Support Supervised Exercise Therapy in Patients With Peripheral Arterial Disease: Study Protocol for a Randomized Controlled Pilot Trial. JMIR Res Protoc. 2019 Jun 26;8(6):e13651. doi: 10.2196/13651. PMID 31244477
- [Derived] Paldan K, Steinmetz M, Simanovski J, Rammos C, Ullrich G, Janosi RA, Moebus S, Rassaf T, Lortz J. Supervised Exercise Therapy Using Mobile Health Technology in Patients With Peripheral Arterial Disease: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Aug 16;9(8):e24214. doi: 10.2196/24214. PMID 34398800

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT04947228/SAP_000.pdf